CLINICAL TRIAL: NCT01793012
Title: Drug Monitoring of Antibiotics in Critical Care Patients
Acronym: DRAK
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Michael Zoller MD, senior physician, Ludwig-Maximilians - University of Munich
Other Study IDs: MUC 428-12; DRKS00004426 (Other: German clinical trials register)
Record Dates: First submitted 2013-01-24; First posted 2013-02-15 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: ARDS; Sepsis
Keywords: therapeutic drug monitoring; antibiotics; inflammation parameters; critically ill patients; septicaemia; intensive care unit
MeSH Terms: conditions — Sepsis; Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- critically ill intensive care patients: Treatment with one or more of the following antibiotics: piperacillin/tazobactam, cefepime, meropenem, ciprofloxacin, linezolid, colistin

SUMMARY:
Infections are critical factors for the survival of critically ill patients. A broad, high-dose and early initial therapy of antibiotics is of particular relevance.

A serious problem is the high variability of antibiotic serum concentrations after administration of antibiotics in patients of the critical care units. This may result in the risk of underdosage with possible ineffective therapeutic levels as well as in the risk of overdosage with possible adverse and toxic effects. The goal of this study is to determine antibiotic concentrations in blood and to evaluate concentrations with the course of the therapy. The measurement of antibiotic concentrations in blood may allow an individual adaption of the dose in future.

100 - 200 patients will be included in this study. Only critically ill patients of the ICU of the Department of Anaesthesiology will be included that receive one or more of the following antibiotics: piperacillin/tazobactam, cefepime, meropenem, ciprofloxacin, linezolid, and colistin.

DETAILED DESCRIPTION:
Substantial variations of serum concentrations of different antibiotics with partly insufficient levels have been observed in critically ill patients. The high variabilities between the pharmacokinetic parameters in different patients argue for a therapeutic drug monitoring (TDM) in intensive care units. TDM may lower the risk of overdosage with possible adverse and toxic effects as well as the risk of underdosage with possible insufficient therapeutic effects and development of antibiotic resistance. The aim of this study is to evaluate variabilities of pharmacokinetic parameters of different widely used antibiotics and to correlate them with clinical and laboratory parameters. Therefore, numerous clinical and laboratory parameters including serum, urine and dialysate concentrations of 6 different antibiotics will be determined in 100 - 200 critically ill patients of the Department of Anaesthesiology, University Hospital of Munich. Laboratory parameters (e.g. inflammatory parameters) will be quantified by facilities of the Institute of Laboratory Medicine, University Hospital of Munich. Concentrations of antibiotics will be determined by liquid chromatography-mass spectrometry (LC-MS/MS). We expect that correlations between antibiotic serum concentrations and clinical and laboratory outcome parameters will be found.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalisation in the critical care unit of the Department of Anaesthesiology of the University Hospital of Munich
2. Presence of infection by clinical assessment
3. Treatment of the patients with one or more of the following antibiotics: piperacillin/tazobactam, cefepime, meropenem, ciprofloxacin, linezolid, colistin
4. Bolus administration of selected antibiotics
5. Valid informed consent subscribed by the patient or by his or her legal guardian or - if only a provisional guardian is defined - by the provisional guardian.

Exclusion Criteria:

1. Prophylactic antibiotics without clinical assessment for the presence of infection
2. Planned shorter hospital stay than 4 days
3. Administration of the selected antibiotic 14 days to 48 hours before the begin of the study
4. Only a single dose of an antibiotic per day
5. Subsequent withdrawal of the participation in the study by the patient or the guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalisation in the critical care unit of the Department of Anaesthesiology of the University Hospital of Munich
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Variability of antibiotic serum concentrations in critically ill patients | 2 Years
  The primary goal of this study is to evaluate the variability of antibiotic serum concentrations in critically ill patients. In total, serum concentrations of 6 different antibiotics (piperacillin/tazobactam, cefepime, meropenem, ciprofloxacin, linezolid, and colistin) in 100-200 patients of the ICU will be determined by liquid chromatography mass spectrometry.

SECONDARY OUTCOMES:
correlate these serum concentrations with clinical and laboratory outcome Correlate serum concentrations with clinical and laboratory outcome parameters | 2 Years
  Moreover, we will evaluate if antibiotic serum concentrations differ between the different diseases (e.g. ARDS, sepsis) and the different therapies (e.g. different transplantation types (liver,lung) patients with and without renal replacement therapy).
  Correlation between antibiotics serum concentrations and Apache II score / SOFA score. Correlation between antibiotics serum concentrations and CRP, procalcitonin, interleukin-6.
  Finally minimal inhibitory concentrations (MIC) of antibiotics will be documented in case of detection of pathogens.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Zwissler, Prof.Dr.med., Study Director — Department of Anaesthesiology of the University Hospital of Munich; Daniel Teupser, Prof.Dr.med., Study Director — Institute of Laboratory Medicine of the University Hospital of Munich; Johannes Zander, Dr. med., Principal Investigator — Institute of Laboratory Medicine of the University Hospital of Munich; Michael Zoller, Dr. med., Principal Investigator — Department of Anaesthesiology of the University Hospital of Munich; Lorenz Frey, Dr. med., Study Chair — Department of Anaesthesiology of the University Hospital of Munich; Michael Vogeser, Prof.Dr.med., Study Chair — Institute of Laboratory Medicine of the University Hospital of Munich; Mathias Bruegel, Dr. med., Study Chair — Institute of Laboratory Medicine of the University Hospital of Munich; Lesca Holdt, Dr.rer.nat., Study Chair — Institute of Laboratory Medicine of the University Hospital of Munich
Locations (1):
- Department of Anaesthesiology of the University Hospital of Munich, Munich, Germany

REFERENCES:
- [Derived] Bilal M, Zoller M, Fuhr U, Jaehde U, Ullah S, Liebchen U, Busker S, Zander J, Babouee Flury B, Taubert M. Cefepime Population Pharmacokinetics, Antibacterial Target Attainment, and Estimated Probability of Neurotoxicity in Critically Ill Patients. Antimicrob Agents Chemother. 2023 Jul 18;67(7):e0030923. doi: 10.1128/aac.00309-23. Epub 2023 Jun 27. PMID 37366614
- [Derived] Ehmann L, Zoller M, Minichmayr IK, Scharf C, Maier B, Schmitt MV, Hartung N, Huisinga W, Vogeser M, Frey L, Zander J, Kloft C. Role of renal function in risk assessment of target non-attainment after standard dosing of meropenem in critically ill patients: a prospective observational study. Crit Care. 2017 Oct 21;21(1):263. doi: 10.1186/s13054-017-1829-4. PMID 29058601
- [Derived] Taubert M, Zoller M, Maier B, Frechen S, Scharf C, Holdt LM, Frey L, Vogeser M, Fuhr U, Zander J. Predictors of Inadequate Linezolid Concentrations after Standard Dosing in Critically Ill Patients. Antimicrob Agents Chemother. 2016 Aug 22;60(9):5254-61. doi: 10.1128/AAC.00356-16. Print 2016 Sep. PMID 27324768
- [Derived] Zander J, Dobbeler G, Nagel D, Maier B, Scharf C, Huseyn-Zada M, Jung J, Frey L, Vogeser M, Zoller M. Piperacillin concentration in relation to therapeutic range in critically ill patients--a prospective observational study. Crit Care. 2016 Apr 4;20:79. doi: 10.1186/s13054-016-1255-z. PMID 27039986
- [Derived] Zoller M, Maier B, Hornuss C, Neugebauer C, Dobbeler G, Nagel D, Holdt LM, Bruegel M, Weig T, Grabein B, Frey L, Teupser D, Vogeser M, Zander J. Variability of linezolid concentrations after standard dosing in critically ill patients: a prospective observational study. Crit Care. 2014 Jul 10;18(4):R148. doi: 10.1186/cc13984. PMID 25011656